CLINICAL TRIAL: NCT01430624
Title: Prevention of Postrape Drug Abuse: Replication Study
Brief Title: Prevention of Post Sexual Assault Stress
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01DA023099 (NIH); R01DA023099 (NIH)
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Drug Use; Drug Abuse; Posttraumatic Stress Disorder
Keywords: Rape; Secondary prevention; Intervention
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PPRS video (Experimental): Prevention of post sexual assault stress
  Interventions: Behavioral: PPRS
- PIRI video (Active Comparator): Pleasant imagery and relaxation instruction
  Interventions: Behavioral: PIRI
- Standard care (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: PPRS — Video including information psychoeducation and modeling of adaptive behavioral coping strategies for use post-assault. Shown at time of post assault medical exam.
  Arms: PPRS video
Behavioral: PIRI — Video containing pleasant imagery and relaxation instruction information. Shown at time of post assault medical exam.
  Arms: PIRI video

SUMMARY:
The purpose of this study is to evaluate whether a brief intervention in video format, that includes education about reactions to assault and modeling of adaptive coping strategies, designed to reduce post assault drug use or abuse and PTSD and shown to recent victims of sexual assault at the time of receipt of post assault medical care is associated with better post-assault outcomes as compared to a comparable length video that includes pleasant imagery and relaxation instruction or standard care.

DETAILED DESCRIPTION:
Post assault outcomes include coping behaviors and PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Seeking medical care after recent sexual assault

Exclusion Criteria:

* Active psychosis Active suicidality Cognitive impairment Non-English speaking Severe injury

Ages: 15 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2009-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Resnick, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Center, Minneapolis, Minnesota

REFERENCES:
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783
- [Derived] Walsh K, Gilmore AK, Jaffe AE, Frazier P, Ledray L, Acierno R, Ruggiero KJ, Kilpatrick DG, Resnick HS. A preliminary examination of sexual and physical victimization 6 months after recent rape. Arch Womens Ment Health. 2023 Aug;26(4):495-501. doi: 10.1007/s00737-023-01335-y. Epub 2023 Jun 8. PMID 37286883
- [Derived] Walsh K, Gilmore AK, Schumacher JA, Coffey SF, Frazier PA, Ledray L, Acierno R, Ruggiero KJ, Kilpatrick DG, Resnick HS. Post-sexual assault cigarette smoking: Findings from a randomized clinical trial of a video-based intervention. Addict Behav. 2020 Jan;100:106121. doi: 10.1016/j.addbeh.2019.106121. Epub 2019 Sep 5. PMID 31622944
- [Derived] Gilmore AK, Walsh K, Frazier P, Ledray L, Acierno R, Ruggiero KJ, Kilpatrick DG, Resnick HS. Prescription Opioid Misuse After a Recent Sexual Assault: A Randomized Clinical Trial of a Video Intervention. Am J Addict. 2019 Sep;28(5):376-381. doi: 10.1111/ajad.12922. Epub 2019 Jun 26. PMID 31242340

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PPRS Video | PIRI Video | Standard Care
Started | 82 (Initial potential eligible screened enrolled) | 82 | 81
Eligible Baseline Completes | 77 | 77 | 79
Completed | 54 (Completed one or more follow-ups) | 48 (Completed one or more follow-ups) | 52 (Completed one or more follow-ups)
Not Completed | 28 | 34 | 29
Not completed — Lost to Follow-up | 23 | 29 | 27
Not completed — technical or eligibility | 5 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- PPRS (Completing Baseline): Prevention of Post-Sexual Assault Stress
- PIRI (Completing Baseline): Pleasant Imagery and Relaxation Instruction
- Standard Care (Completing Baseline): Standard Care Condition completing baseline
- Total: Total of all reporting groups
Arm/Group | PPRS (Completing Baseline) | PIRI (Completing Baseline) | Standard Care (Completing Baseline) | Total
Number analyzed (Participants) | 77 | 77 | 79 | 233
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 5 | 2 | 10
  Between 18 and 65 years | 74 | 72 | 77 | 223
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.79 (8.22) | 27.99 (10.77) | 27.52 (10.01) | 27.43 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 77 | 79 | 233
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 77 | 77 | 79 | 233

OUTCOME MEASURES:

1. Primary Outcome: Drug Abuse Screening Test (DAST-10)
Description: total possible scores range from 0 - 10 with higher scores indicating poor functioning, post assault at 6 months
Time Frame: 6 months
Population: Only includes participants with complete scale data at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PPRS Video | PIRI Video | Standard Care
Number analyzed (Participants) | 34 | 39 | 39
units on a scale | 1.97 (2.65) | 2.03 (2.85) | 1.18 (1.62)
Statistical Analysis 1: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .24, ANOVA — 6 month follow-up comparison; df 2, 109

2. Primary Outcome: Alcohol Use Disorders Identification Test (AUDIT)
Description: Total scores range from 0 - 40 with higher scores indicating greater problem severity, post assault at 6 months
Time Frame: 6 months
Population: Includes only participants with full scale score information at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PPRS Video | PIRI Video | Standard Care
Number analyzed (Participants) | 33 | 40 | 41
units on a scale | 7.21 (8.73) | 7.53 (9.69) | 8.15 (7.42)
Statistical Analysis 1: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .89, ANOVA — 6 month follow-up comparison; df = 2, 111

3. Primary Outcome: Cigarettes (Estimated Number)
Description: quantity in 14 days prior to 6 week, 3 month and 6 month follow-up
Time Frame: 14 days preceding 6 week, 3 month and 6 month follow-up
Population: 1 participant missing 6 week cigarette smoking information
Measure: Mean (Standard Error); unit: cigarettes
Groups:
- PPRS: Prevention of Post-Sexual Assault Stress
- PIRI: Pleasant Imagery and Relaxation Condition
- SC Condition: Standard Care Completing Follow-up
Arm/Group | PPRS | PIRI | SC Condition
Number analyzed (Participants) | 53 | 48 | 52
cigarettes
  6 Week (n = 53, 48, 52) | 49.94 (80.19) | 87.29 (141.20) | 118.04 (114.94)
  3 Month (n = 48, 44, 43) | 54.63 (121.22) | 67.73 (129.01) | 84.47 (100.54)
  6 Month (n = 38, 41, 42) | 42.68 (76.78) | 71.71 (126.15) | 84.64 (92.67)
Statistical Analysis 1: Comparison: PPRS vs PIRI vs SC Condition; Test type: Superiority or Other; p = .01, ANOVA — 6 week comparison; df = 2, 150
Statistical Analysis 2: Comparison: PPRS vs PIRI vs SC Condition; Test type: Superiority or Other; p = .48, ANOVA — 3 month comparison
Statistical Analysis 3: Comparison: PPRS vs PIRI vs SC Condition; Test type: Superiority or Other; p = .17, ANOVA — 6 month comparison

4. Secondary Outcome: Any Other Illicit Drug Use
Description: Any reported use of cocaine or other illicit drugs other than marijuana in the 14 days prior to follow-up
Time Frame: 14 days prior to 6 week, 3 month, 6 month follow-up
Measure: Number; unit: participants
Arm/Group | PPRS Video | PIRI Video | Standard Care
Number analyzed (Participants) | 54 | 48 | 52
participants
  6 Week (n = 54, 48, 52) | 6 | 0 | 2
  3 Month (n = 48, 42, 43) | 4 | 3 | 2
  6 Month (n = 38, 41, 42) | 4 | 4 | 3
Statistical Analysis 1: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .37, Chi-squared — 6 week comparison; df = 2, 154
Statistical Analysis 2: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .15, Chi-squared — 3 month comparison; df = 2, 135
Statistical Analysis 3: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .87, Chi-squared — 6 month comparison; df = 2, 121

5. Primary Outcome: Amount of Alcohol Use
Description: estimated number of drinks during the 14 days prior to each follow-up assessment
Time Frame: 14 days prior to 6 week, 3 month, 6 month follow-up
Population: 1 participant with missing data at 6 week follow-up
Measure: Mean (Standard Deviation); unit: Drinks
Arm/Group | PPRS Video | PIRI Video | Standard Care
Number analyzed (Participants) | 54 | 48 | 51
Drinks
  6 Week (n = 54, 48, 51) | 15.33 (21.20) | 13.92 (28.17) | 19.90 (43.73)
  3 Month (n = 48, 44, 43) | 8.29 (12.81) | 14.32 (22.47) | 11.49 (15.66)
  6 Month (n = 38, 41, 42) | 10.16 (21.42) | 10.49 (21.58) | 14.60 (22.62)
Statistical Analysis 1: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .63, ANOVA — 6 week comparison; df = 2, 150
Statistical Analysis 2: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .25, ANOVA — 3 month comparison; df = 2, 132
Statistical Analysis 3: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .59, ANOVA — 6 month comparison; df = 2, 118

6. Primary Outcome: Marijuana Use Frequency
Description: Number of days of use within the 14 days prior to follow-up assessment
Time Frame: 14 days prior to 6 week, 3 month, 6 month follow-up
Measure: Mean (Standard Deviation); unit: days of use
Arm/Group | PPRS Video | PIRI Video | Standard Care
Number analyzed (Participants) | 54 | 48 | 52
days of use
  6 Week (n = 54, 48, 52) | 1.98 (3.85) | 2.48 (4.52) | 2.12 (4.42)
  3 Month (n = 48, 44, 43) | 2.75 (4.94) | 1.39 (2.81) | 2.12 (4.28)
  6 Month (n = 38, 41, 42) | 1.03 (2.70) | 1.73 (3.98) | 2.90 (5.40)
Statistical Analysis 1: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .83, ANOVA — 6 week comparison; df = 2, 151
Statistical Analysis 2: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .29, ANOVA — 3 month comparison; df = 2, 132
Statistical Analysis 3: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .13, ANOVA — 6 month comparison; df = 2, 118

7. Secondary Outcome: Non-medical Use of Prescription Drugs Frequency
Description: Number of days of use within the 14 days prior to follow-up assessment
Time Frame: 14 days prior to 6 week, 3 month, 6 month follow-up
Population: 2 participants had missing data at 6 month follow-up
Measure: Mean (Standard Deviation); unit: days of use
Arm/Group | PPRS Video | PIRI Video | Standard Care
Number analyzed (Participants) | 54 | 48 | 52
days of use
  6 Week (n = 54, 48, 52) | 1.56 (3.96) | .08 (.35) | .54 (1.60)
  3 Month (n = 48, 44, 43) | .81 (2.57) | .75 (2.63) | .16 (.62)
  6 Month (n = 38, 40, 41) | .61 (2.39) | .40 (1.19) | .10 (.63)
Statistical Analysis 1: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .012, ANOVA — 6 week comparison; df = 2, 151
Statistical Analysis 2: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .31, ANOVA — 3 month comparison; df = 2, 132
Statistical Analysis 3: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .35, ANOVA — 6 month comparison; df = 2,116

8. Secondary Outcome: PTSD Symptom Scale Self-Report (PSS-SR)
Description: Total scores range from 0 to 51 with higher scores indicating greater frequency of symptoms, Measure of PTSD symptoms.
Time Frame: 2 weeks prior to 6 week, 3 month, 6 month followup
Population: Only includes those with complete scale score information
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard Care: Treatment as usual which included standard care
Arm/Group | PPRS Video | PIRI Video | Standard Care
Number analyzed (Participants) | 52 | 43 | 49
units on a scale
  6 Week (n = 52, 43, 49) | 26.98 (10.42) | 29.07 (11.48) | 24.49 (11.63)
  3 Month (n = 45, 42, 43) | 23.98 (11.09) | 23.33 (13.03) | 21.70 (12.56)
  6 Month (n = 35, 37, 41) | 17.66 (11.83) | 21.65 (12.80) | 19.83 (12.47)
Statistical Analysis 1: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .15, ANOVA — 6 week comparison; df = 2, 141
Statistical Analysis 2: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .67, ANOVA — 3 month comparison; df = 2, 127
Statistical Analysis 3: Comparison: PPRS Video vs PIRI Video vs Standard Care; Test type: Superiority or Other; p = .40, ANOVA — 6 month comparison; df = 2, 110

ADVERSE EVENTS:
Time Frame: 6 months
Description: Cause of death and cause of hospitalization unknown
Groups:
- PIRI: Pleasant Imagery and Relaxation Instruction
- Standard Care Condition: Standard Care Condition
Arm/Group | PPRS | PIRI | Standard Care Condition
Serious Adverse Events (participants affected / at risk) | 2/82 | 0/82 | 0/81
Other Adverse Events (participants affected / at risk) | 0/82 | 0/82 | 0/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PPRS (N=82) | PIRI (N=82) | Standard Care Condition (N=81)
death (General disorders) | 1 (1) | 0 (0) | 0 (0) — unanticipated, unlikely/unrelated to study - no information about cause, identified over course of study and not related to study procedures
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Unlikely/unrelated to study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No